CLINICAL TRIAL: NCT03909646
Title: Surgical Excision Versus Photodynamic Therapy and Topical 5-fluorouracil in Treatment of Bowen's Disease: a Multicenter Randomized Controlled Trial
Brief Title: Surgical Excision Versus Photodynamic Therapy and Topical 5-fluorouracil in Treatment of Bowen's Disease
Acronym: BOWTIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 67545
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Bowen's Disease
MeSH Terms: conditions — Bowen's Disease | interventions — methyl 5-aminolevulinate; Myelin and Lymphocyte-Associated Proteolipid Proteins; Fluorouracil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Surgical excision (Active Comparator): Standard surgical excision with 5 mm safety margin
  Interventions: Other: Surgical excision
- Photodynamic therapy (Active Comparator): PDT with application of methyl aminolevulinate (MAL) cream followed by two illuminations with a one-week interval
  Interventions: Drug: Methyl Aminolevulinate (Mal) for Topical Administration, 16.8%, 1 Gram
- 5% 5-Fluorouracil (Active Comparator): 5FU cream, which has to be applied by the patient twice daily for 4 weeks.
  Interventions: Drug: 5Fluorouracil

INTERVENTIONS:
Drug: Methyl Aminolevulinate (Mal) for Topical Administration, 16.8%, 1 Gram — A layer of methylaminolevulinc acid 160 mg/g cream (about 1 mm thick) is applied to the lesion, with a clinical margin of 5-10 mm surrounding of normal skin and then covered by an occlusive dressing. After 3 hours the occlusive dressing will be removed and the area is illuminated with Omnilux or Actilite (Galderma). After PDT the treatment site is covered again with the above mentioned occlusive dressings during 48 hours. Treatment is performed by an authorized nurse in the hospital. Two sessions should be administered with an interval of one week between sessions.
  Other Names: Metvix
  Arms: Photodynamic therapy
Drug: 5Fluorouracil — 5-FU is applied on the treatment area by the patient in a thin layer twice daily during 4 weeks.
  Other Names: Efudix
  Arms: 5% 5-Fluorouracil
Other: Surgical excision — Local anesthesia with lidocain 1% (1-2ml) will be used before performing standard surgical excision with 5 mm safety margin followed by routine histological examination. The skin will be closed using cutaneous sutures, which will be removed after 1-2 weeks. The surgical excision will take place in the hospital by the treating physician
  Arms: Surgical excision

SUMMARY:
There is limited quality research on the effectiveness of treatments in Bowen's disease (BD). Patient and lesion characteristics, patient preferences and costs should be considered when choosing therapy. Surgical excision (SE), photodynamic therapy (PDT) and 5-fluorouracil (5FU) are mentioned as treatment options in guidelines. However no clear and evidence based recommendations are made in terms of effectiveness.

Objective: The aim of this study is 1) to evaluate the (cost)effectiveness of 5FU and PDT compared to SE in BD and 2) to compare the effectiveness of 5FU with that of PDT. With a better understanding of the (cost)effectiveness of alternative treatment options, the investigators will supply the necessary evidence for national and international guidelines, to achieve more uniformity in treatment of BD.

Study design: Randomized controlled non-inferiority multicenter trial. Study population: Patients ≥18 years, with a histological proven primary lesion of Bowen's disease, visiting Maastricht University Medical Centre, Catharina hospital Eindhoven, VieCuri MC Venlo or Zuyderland Medical Centre Heerlen.

Intervention: One group undergoes SE with a 5mm safety margin followed by routine histological examination. The other group receives PDT with application of methyl aminolevulinate (MAL) cream followed by two illuminations with a one-week interval. The third group receives 5FU cream, which has to be applied by the patient twice daily for 4 weeks.

Main study parameters/endpoints: The primary outcome is the proportion of patients with sustained clearance at 12 months post-treatment. Secondary outcomes are proportion of patients with clearance at 3 months, the long-term probability of sustained clearance, cost-effectiveness, patient satisfaction, patient preferences, compliance, side effects and cosmetic outcome. Post-treatment, patients will be asked to answer a short questionnaire regarding side effects, experience with the treatment and satisfaction.

DETAILED DESCRIPTION:
This is a multicenter randomized controlled non-inferiority trial, conducted in one academic and three non-academic hospitals. A multicenter approach (academic and non-academic centers) increases the generalizability of the study results. The study takes place at the dermatology department of Maastricht University Medical Centre (MUMC+), Catharina hospital Eindhoven, VieCuri Medical Centre Venlo and Zuyderland Medical Centre Heerlen.

A non-inferiority design was chosen because although the noninvasive treatments are expected to be somewhat less effective in terms of remaining free of recurrence, there are other benefits such as higher patient satisfaction, patient preferences and better cosmetic outcome. It should be noted that BD is a noninvasive disease and recurrences can be treated with surgical excision without compromising the patient's health.

After giving permission and signing the informed consent form, eligible patients will be randomly assigned to one of three treatment groups: 1) PDT, 2) 5% 5FU cream, 3) surgical excision. All interventions are part of regular care. For the treatment of BD 5% 5FU cream (Efudix®) has been approved by the European Medicines Agency (EMA).

The coordinating investigator who is not blinded to the randomized treatment will prescribe the 5FU cream or give orders to plan PDT or excision and provide patients with further information. The supervising dermatologist will be blinded to treatment allocation, and will be asked to assess outcome measures such as clearance and cosmetic evaluation. Relevant baseline characteristics will be registered (e.g. prior history of skin cancer, age, gender, use of immunosuppressant medication in history, prior treatments for non-melanoma skin cancer), dermatological description of the lesion, size and localization of the lesion and the histological tumour thickness. The presence of other lesions, besides the target lesion, and their treatment will be recorded

The primary outcome will be the proportion of patients with sustained clearance at 12 months follow-up after the end of treatment. Secondary outcomes will be the proportion of patients with clearance at 3 months, the long-term probability of sustained clearance, cost-effectiveness, patient satisfaction, compliance, side effects and cosmetic outcome.

Residual tumour at 3 months follow-up and recurrent tumour at 12 months follow-up is considered as treatment failure and will be treated with surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years
* Histologically proven primary Bowen's disease
* Lesions ≥ 4mm and ≤ 40mm in diameter
* Fitzpatrick skin type I-IV
* Female in child bearing potential should be using contraceptive measures, during and till 3 months post-treatment

Exclusion Criteria:

* Bowen's Disease located at ears, periocular, nail unit or periungual tissue, nose, genital and mucous membranes
* High clinical suspicion of invasive SCC
* Interfering treatment of other (N)MSC in target area
* Not able to self-apply cream on lesions located on the back or other difficult to reach locations
* Pregnancy
* Breastfeeding
* Allergy to study drugs
* Genetic skin cancer disorders
* Not understanding Dutch language
* Porphyria
* Not able to give informed consent
* Immuno-compromised status
* Use of systemic retinoid in the past 3 months
* Use of immunosuppressant drugs in the past 3 months and / or at time of treatment (such as oral glucocorticoids, cytostatic, antibodies, drug acting on immunophilins, in-terferon, opioids, TNF binding proteins, MMF, biologic agents). Inhalation corticoster-oids / nasal corticosteroids are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-27 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Sustained clearance (no residue, recurrence nor progression) | 12 months post-treatment
  The main study endpoint is the proportion of patients with sustained clearance (no residue, recurrence nor progression) 12 months post-treatment.

SECONDARY OUTCOMES:
the proportion of patients with clearance at 3 months post-treatment, the long-term probability of sustained clearance, cost-effectiveness, patient satisfaction, patient preferences, compliance, side effects and cosmetic outcome. | 3 months and at least 3 years post-treatment
  the proportion of patients with clearance at 3 months post-treatment, the long-term probability of sustained clearance, cost-effectiveness, patient satisfaction, patient preferences, compliance, side effects and cosmetic outcome.
  Long-term is defined as at least 3 years post-treatment. All patients will be invited for the long-term follow-up visit at least 3 years after finishing treatment, with the last patient finishing treatment at April 16th 2021.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Mosterd, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holterhues C, Vries Ed, Louwman MW, Koljenovic S, Nijsten T. Incidence and trends of cutaneous malignancies in the Netherlands, 1989-2005. J Invest Dermatol. 2010 Jul;130(7):1807-12. doi: 10.1038/jid.2010.58. Epub 2010 Mar 25. PMID 20336085
- [Background] Arlette JP, Trotter MJ. Squamous cell carcinoma in situ of the skin: history, presentation, biology and treatment. Australas J Dermatol. 2004 Feb;45(1):1-9; quiz 10. doi: 10.1111/j.1440-0960.2004.00025.x. PMID 14961900
- [Background] Bowen JT. Centennial paper. May 1912 (J Cutan Dis Syph 1912;30:241-255). Precancerous dermatoses: a study of two cases of chronic atypical epithelial proliferation. By John T. Bowen, M.D., Boston. Arch Dermatol. 1983 Mar;119(3):243-60. No abstract available. PMID 6297414
- [Background] Shimizu I, Cruz A, Chang KH, Dufresne RG. Treatment of squamous cell carcinoma in situ: a review. Dermatol Surg. 2011 Oct;37(10):1394-411. doi: 10.1111/j.1524-4725.2011.02088.x. Epub 2011 Jul 18. PMID 21767324
- [Background] Kao GF. Carcinoma arising in Bowen's disease. Arch Dermatol. 1986 Oct;122(10):1124-6. No abstract available. PMID 3767398
- [Background] PETERKA ES, LYNCH FW, GOLTZ RW. An association between Bowen's disease and internal cancer. Arch Dermatol. 1961 Oct;84:623-9. doi: 10.1001/archderm.1961.01580160087015. No abstract available. PMID 14485715
- [Background] Bichakjian CK, Olencki T, Aasi SZ, Alam M, Andersen JS, Berg D, Bowen GM, Cheney RT, Daniels GA, Glass LF, Grekin RC, Grossman K, Higgins SA, Ho AL, Lewis KD, Lydiatt DD, Nehal KS, Nghiem P, Olsen EA, Schmults CD, Sekulic A, Shaha AR, Thorstad WL, Tuli M, Urist MM, Wang TS, Wong SL, Zic JA, Hoffmann KG, Engh A. Basal Cell Skin Cancer, Version 1.2016, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2016 May;14(5):574-97. doi: 10.6004/jnccn.2016.0065. PMID 27160235
- [Background] Bath-Hextall FJ, Matin RN, Wilkinson D, Leonardi-Bee J. Interventions for cutaneous Bowen's disease. Cochrane Database Syst Rev. 2013 Jun 24;2013(6):CD007281. doi: 10.1002/14651858.CD007281.pub2. PMID 23794286
- [Background] Bonerandi JJ, Beauvillain C, Caquant L, Chassagne JF, Chaussade V, Clavere P, Desouches C, Garnier F, Grolleau JL, Grossin M, Jourdain A, Lemonnier JY, Maillard H, Ortonne N, Rio E, Simon E, Sei JF, Grob JJ, Martin L; French Dermatology Recommendations Association (aRED). Guidelines for the diagnosis and treatment of cutaneous squamous cell carcinoma and precursor lesions. J Eur Acad Dermatol Venereol. 2011 Dec;25 Suppl 5:1-51. doi: 10.1111/j.1468-3083.2011.04296.x. No abstract available. PMID 22070399
- [Background] Hansen JP, Drake AL, Walling HW. Bowen's Disease: a four-year retrospective review of epidemiology and treatment at a university center. Dermatol Surg. 2008 Jul;34(7):878-83. doi: 10.1111/j.1524-4725.2008.34172.x. PMID 18363722
- [Background] Morley GL, Matthews JH, Verpetinske I, Thom GA. A Comparative Study Examining the Management of Bowen's Disease in the United Kingdom and Australia. Dermatol Res Pract. 2015;2015:421460. doi: 10.1155/2015/421460. Epub 2015 Sep 9. PMID 26442118
- [Background] Morton CA, Birnie AJ, Eedy DJ. British Association of Dermatologists' guidelines for the management of squamous cell carcinoma in situ (Bowen's disease) 2014. Br J Dermatol. 2014 Feb;170(2):245-60. doi: 10.1111/bjd.12766. No abstract available. PMID 24313974
- [Background] Overmark M, Koskenmies S, Pitkanen S. A Retrospective Study of Treatment of Squamous Cell Carcinoma In situ. Acta Derm Venereol. 2016 Jan;96(1):64-7. doi: 10.2340/00015555-2175. PMID 26073523
- [Background] Szeimies RM, Karrer S, Backer H. [Therapeutic options for epithelial skin tumors. Actinic keratoses, Bowen disease, squamous cell carcinoma, and basal cell carcinoma]. Hautarzt. 2005 May;56(5):430-40. doi: 10.1007/s00105-005-0950-5. German. PMID 15815888
- [Background] Westers-Attema A, van den Heijkant F, Lohman BG, Nelemans PJ, Winnepenninckx V, Kelleners-Smeets NW, Mosterd K. Bowen's disease: A six-year retrospective study of treatment with emphasis on resection margins. Acta Derm Venereol. 2014 Jul;94(4):431-5. doi: 10.2340/00015555-1771. PMID 24337161
- [Background] Jansen MH, Appelen D, Nelemans PJ, Winnepenninckx VJ, Kelleners-Smeets NWJ, Mosterd K. Bowen's Disease: Long-term Results of Treatment with 5-Fluorouracil Cream, Photodynamic Therapy or Surgical Excision. Acta Derm Venereol. 2018 Jan 12;98(1):114-115. doi: 10.2340/00015555-2777. No abstract available. PMID 29135015
- [Background] Arits AH, Mosterd K, Essers BA, Spoorenberg E, Sommer A, De Rooij MJ, van Pelt HP, Quaedvlieg PJ, Krekels GA, van Neer PA, Rijzewijk JJ, van Geest AJ, Steijlen PM, Nelemans PJ, Kelleners-Smeets NW. Photodynamic therapy versus topical imiquimod versus topical fluorouracil for treatment of superficial basal-cell carcinoma: a single blind, non-inferiority, randomised controlled trial. Lancet Oncol. 2013 Jun;14(7):647-54. doi: 10.1016/S1470-2045(13)70143-8. Epub 2013 May 15. PMID 23683751
- [Background] Morton CA, McKenna KE, Rhodes LE; British Association of Dermatologists Therapy Guidelines and Audit Subcommittee and the British Photodermatology Group. Guidelines for topical photodynamic therapy: update. Br J Dermatol. 2008 Dec;159(6):1245-66. doi: 10.1111/j.1365-2133.2008.08882.x. Epub 2008 Oct 13. PMID 18945319
- [Background] M Versteegh M, M Vermeulen K, M A A Evers S, de Wit GA, Prenger R, A Stolk E. Dutch Tariff for the Five-Level Version of EQ-5D. Value Health. 2016 Jun;19(4):343-52. doi: 10.1016/j.jval.2016.01.003. Epub 2016 Mar 30. PMID 27325326
- [Background] Briggs AH, Wonderling DE, Mooney CZ. Pulling cost-effectiveness analysis up by its bootstraps: a non-parametric approach to confidence interval estimation. Health Econ. 1997 Jul-Aug;6(4):327-40. doi: 10.1002/(sici)1099-1050(199707)6:43.0.co;2-w. PMID 9285227
- [Derived] Ahmady S, van Riel CAM, Kelleners-Smeets NWJ, Mosterd K, Essers BAB. Cost-Effectiveness of Photodynamic Therapy and 5-Fluorouracil Cream versus Surgical Excision in Treatment of Bowen's Disease: A Trial-Based Economic Evaluation. Dermatology. 2025;241(5-6):489-498. doi: 10.1159/000548431. Epub 2025 Sep 11. PMID 40934140